CLINICAL TRIAL: NCT01739686
Title: Collaborative Care to Alleviate Symptoms and Adjust to Illness in Chronic Heart Failure (CASA) Trial
Acronym: CASA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Research Institute (Other)
Collaborators: VA Eastern Colorado Health Care System (U.S. Federal Agency); University of Colorado, Denver (Other); Denver Health Medical Center (Other); University of Iowa (Other)
Responsible Party: Principal Investigator, David Bekelman, M.D., Associate Professor of Medicine, Denver Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5R01NR013422-02 (NIH); 11-0969 (Other: Colorado Multiple Institutional Review Board (COMIRB))
Record Dates: First submitted 2012-11-16; First posted 2012-12-03 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Chronic Heart Failure
Keywords: Quality of Life; Symptoms; Palliative care; Symptom management; Disease management; Health delivery

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CASA Intervention (Experimental): The CASA (Collaborative Care to Alleviate Symptoms and Adjust to Illness) intervention includes 3 components:
  * A nurse (RN) follows structured algorithms to help patients with symptoms, specifically breathlessness, fatigue, pain, and depression.
  * A social worker provides structured counseling targeting adjustment to illness and depression if present.
  * A collaborative care model of care delivery, in which the nurse and social worker meet weekly with a primary care provider, cardiologist and palliative care specialist. This team makes medical recommendations to the intervention subjects' providers and supervises the nurse and social worker.
  Most of the nurse and social worker visits are by phone.
  Interventions: Other: CASA Intervention
- Usual Care (No Intervention): Patients in the control group will continue to receive care at the discretion of their providers, which may include referral to cardiology, palliative care, or mental health. If patients self-report depression on baseline surveys, this information will be given to their provider, and patients will be given resources. Patients will have the same amount of interaction with research assistants as the intervention patients, completing questionnaires and participating in study visits at the same frequency.

INTERVENTIONS:
Other: CASA Intervention — CASA Intervention
  The CASA (Collaborative Care to Alleviate Symptoms and Adjust to Illness) intervention includes 3 components:
  A nurse (RN) follows structured algorithms to help patients with symptoms, specifically breathlessness, fatigue, pain, and depression.
  A social worker provides structured counseling targeting adjustment to illness and depression if present.
  A collaborative care model of care delivery, in which the nurse and social worker meet weekly with a primary care provider, cardiologist and palliative care specialist. This team makes medical recommendations to the intervention subjects' providers and supervises the nurse and social worker.
  Most of the nurse and social worker visits are by phone.
  Arms: CASA Intervention

SUMMARY:
Chronic heart failure is an important public health problem as it is a leading cause of disability, hospitalization, death, and costs. People who live with advanced chronic heart failure suffer from numerous symptoms that affect their daily lives. The investigators are conducting a randomized clinical trial to evaluate a symptom management and psychosocial care intervention to improve health status (symptom burden, functioning, and quality of life). The results will be directly relevant to patients and families who suffer with this illness, as well as to providers, payers, and other researchers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or older
* Able to read and understand English
* Consistent access to a telephone
* Patients have a primary care or other provider who is willing to facilitate intervention medical recommendations
* A diagnosis of heart failure with at least one of the following:

[hospitalization primarily for heart failure in the year prior (including current); taking at least 20 mg oral furosemide (or equivalent) daily in a single or divided dose; Brain natriuretic peptide(BNP) ≥ 100 or N-terminal prohormone of brain natriuretic peptide(NT-proBNP) ≥ 500; EF≤40%]

* Report a low health status (KCCQ-SF≤70)
* Bothered by at least one target symptom:

[Pain; Depression; Fatigue; Breathlessness]

Exclusion Criteria:

* Previous diagnosis of dementia
* Active substance abuse or dependence, defined by either a diagnosis of abuse or dependence or an AUDIT-C ≥ 8, or self-reported substance abuse in the past 3 months
* Comorbid metastatic cancer
* Nursing home resident
* Heart Transplant recipient
* LVAD recipient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Difference in Kansas City Cardiomyopathy Questionnaire (KCCQ) overall score | 6 months
  The KCCQ is a self-administered questionnaire that measures heart failure-specific health status. The KCCQ is reliable, sensitive to clinical change, and predicts hospitalization and mortality. The study will test whether there is a difference in KCCQ overall score between the intervention and control groups at 6 months.

SECONDARY OUTCOMES:
Difference in Patient Health Questionnaire-9 (PHQ-9) score | 6 months
  The PHQ-9 is a 9-item valid and reliable instrument that provides a continuous measure of depressive symptoms and is 88% sensitive and specific for a diagnosis of major depressive disorder. The PHQ-9 was developed in medically-ill outpatients, including patients with heart failure.
Difference in symptom distress, measured using the General Symptom Distress Scale | 6 months
  The General Symptom Distress Scale (GSDS)includes a measure of overall symptom distress and ability to manage symptoms.
Difference in Self-care of Heart Failure Index (SCHFI) | 12 months
  The SCHFI is a valid and reliable 22-item self-report measure of self-care that includes three self-care scales: maintenance, management, and confidence
Difference in Satisfaction with Healthcare | 6 months
Difference in pain using the PEG | 6 months
  The PEG items assess average pain intensity (P), interference with enjoyment of life (E), and interference with general activity (G).
Change in fatigue using the Patient Reported Outcomes Measurement Information System (PROMIS) fatigue measure | 6 months
Change in Dyspnea | 6 months
  PEG pain measure modified to assess breathlessness
Change in Sheehan Disability Scale | 12 months
  Measure of functioning
Change in Quality of Life at the End of Life (QUAL-E) | 12 months
  The QUAL-E is a valid and reliable self-report measure of several domains, each scored separately, of quality of life in advanced illness. We will use the relationship with health care system, preparation, life completion, and global quality of life sub-scales.

CONTACTS AND LOCATIONS:
Overall Officials: David Bekelman, MD, MPH, Principal Investigator — Denver Research Institute
Locations (3):
- United States (3):
  - University of Colorado Hospital, Aurora, Colorado
  - Denver Health, Denver, Colorado
  - VA Eastern Colorado Health Care System(ECHCS), Denver, Colorado

REFERENCES:
- [Derived] Doyon K, Flint K, Albright K, Bekelman D. Improving Benefit and Reducing Burden of Informal Caregiving for Patients With Heart Failure: A Mixed Methods Study. J Cardiovasc Nurs. 2025 Sep-Oct 01;40(5):406-412. doi: 10.1097/JCN.0000000000001137. Epub 2024 Sep 27. PMID 39348302
- [Derived] Graney BA, Portz JD, Bekelman DB. "I Felt Like I Mattered": Caring is a key ingredient of collaborative care for chronic illness. Chronic Illn. 2024 Sep;20(3):383-394. doi: 10.1177/17423953241264862. Epub 2024 Jul 23. PMID 39043359
- [Derived] Bekelman DB, Allen LA, McBryde CF, Hattler B, Fairclough DL, Havranek EP, Turvey C, Meek PM. Effect of a Collaborative Care Intervention vs Usual Care on Health Status of Patients With Chronic Heart Failure: The CASA Randomized Clinical Trial. JAMA Intern Med. 2018 Apr 1;178(4):511-519. doi: 10.1001/jamainternmed.2017.8667. PMID 29482218
- [Derived] Bekelman DB, Allen LA, Peterson J, Hattler B, Havranek EP, Fairclough DL, McBryde CF, Meek PM. Rationale and study design of a patient-centered intervention to improve health status in chronic heart failure: The Collaborative Care to Alleviate Symptoms and Adjust to Illness (CASA) randomized trial. Contemp Clin Trials. 2016 Nov;51:1-7. doi: 10.1016/j.cct.2016.09.002. Epub 2016 Sep 12. PMID 27634669